CLINICAL TRIAL: NCT04466072
Title: The Correlation Between Gut Microbiome-host Interaction and Ventricular Arrhythmias
Brief Title: Gut Microbiome and Ventricular Arrhythmias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: North Florida Foundation for Research and Education (Other)
Responsible Party: Principal Investigator, Ramil Goel, Clinical Electrophysiologist, Malcolm Randall VAMC, Gainesville, North Florida Foundation for Research and Education
Other Study IDs: IRB202001134
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Gut Microbiome
Keywords: Ventricular arrhythmias; microbiome
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Occult Blood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Stool samples will be collected and analyzed for bacterial DNA analysis to characterize nature and function of microbial flora. Host human DNA may be a contaminant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Ventricular Arrhythmia burden group: Inclusion criteria for all groups:
  * age >18 years-old
  * competent and willing to provide consent
  * presence of implantable cardioverter-defibrillator
  * diagnosis of cardiomyopathy
  * left ventricular ejection fraction of 35% or less as assessed by echocardiogram within 1 year prior to enrollment
  Inclusion criteria for high ventricular arrhythmia burden group:
  • at least one episode of sustained VT/VF or VT/VF requiring ICD therapies within the preceding 3 months as assessed on device interrogation at the time of study enrollment
  Both groups will have stool sample collected for microbial analysis. This is anticipated twice for the high ventricular arrhythmia (VA) burden group. Once at the time of diagnosis of VA and later after the clinically indicated treatment for the VA.
  Interventions: Diagnostic Test: Stool test for microbial analysis
- Control group: Inclusion criteria for all groups:
  * age >18 years-old
  * competent and willing to provide consent
  * presence of implantable cardioverter-defibrillator
  * diagnosis of cardiomyopathy
  * left ventricular ejection fraction of 35% or less as assessed by echocardiogram within 1 year prior to enrollment
  Inclusion criteria for control group:
  • no VT/VF on device interrogation for a period of at least 3 months preceding study enrollment
  Both groups will have stool sample collected for microbial analysis. This is anticipated only once for the control group.
  Interventions: Diagnostic Test: Stool test for microbial analysis

INTERVENTIONS:
Diagnostic Test: Stool test for microbial analysis — Fecal samples will be analyzed by shotgun metagenomics and sample from the high ventricular arrhythmia burden will be compared with those from comparable control patients with low ventricular arrhythmia burden.

SUMMARY:
Ventricular tachycardia and ventricular fibrillation (VT/VF) are the most common causes of sudden cardiac death in patients with diseased hearts. The factors contributing to these deadly arrhythmias are not well understood.

The presence of a wide variety of microbial flora in the human GI tract, particularly colon has been well recognized for a long time. There are also emerging links showing the effect of an intact gut microbiome having effects on left ventricular remodeling after myocardial infarction and hypertension. Gut microbiota has also been associated with outcomes in atrial fibrillation.

There is little available in current literature showing a relationship between gut microbiome characteristics and ventricular arrhythmia burden. The gut microbiome has particularly strong interactions with neuroendocrine and immunologic mediators and has effects on the modulation of the autonomic nervous system. These systems are also hypothesized to influence ventricular arrhythmias. The investigators propose to study the relation and interaction between gut microbiome and ventricular arrhythmogenesis.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: To identify specific gut microbiome characteristics of patients who are prone to clinically significant or high burden of ventricular arrhythmias compared with patients with similar conventional risk factors and low burden of ventricular arrhythmias.

Aim 2: To examine changes that occur in the gut microbiome composition after treatment of ventricular arrhythmias.

Research Plan:

This study will enroll 30 subjects recruited from the electrophysiology device clinic at the VA medical center, who are individuals with underlying cardiomyopathy and prone to ventricular arrhythmias.

Out of this cohort, the investigators will identify 2 groups who have different ventricular arrhythmia burden despite similar conventional clinical factors.

This information regarding ventricular arrhythmia burden will be obtained from device interrogation at the time of recruitment. Our proposal is study and compare the fecal microbial composition of these groups to analyze association with ventricular arrhythmia burden. Patients will provide a fecal sample for analysis at the time of enrollment.

After clinically indicated treatment in the high ventricular arrhythmia group, the investigators will retest fecal samples to assess for changes in characteristics after treatment. This will be done to study changes in the gut microbiome with ventricular arrhythmia in the same individual.

After initial testing of the high burden group, they will undergo treatment aimed at decreasing their burden of arrhythmia, with some combination of anti-arrhythmic drugs, sympathetic blockade, or ventricular tachycardia ablation. After demonstrating a period of 3 months without sustained VT/VF on device interrogation, their fecal samples will be re-analyzed. If a patient continues to have VT/VF requiring intermittent device therapies despite a 6 month period of intensification of therapy, their fecal sample will be re-analyzed after that 6 month timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for all groups:

  * age >18 years-old
  * competent and willing to provide consent
  * presence of implantable cardioverter-defibrillator
  * diagnosis of cardiomyopathy
  * left ventricular ejection fraction of 35% or less as assessed by echocardiogram within 1 year prior to enrollment
* Inclusion criteria for control group:

  • no VT/VF on device interrogation for a period of at least 3 months preceding study enrollment
* Inclusion criteria for high ventricular arrhythmia burden group:

  * at least one episode of sustained VT/VF or VT/VF requiring ICD therapies within the preceding 3 months as assessed on device interrogation at the time of study enrollment

Exclusion Criteria:

* currently pregnant or have been pregnant in the last 6 months
* antibiotic treatment within 5 months of study enrollment (i.e. antibiotic therapy in the two months prior to the 3-month period of analysis for VT/VF)
* chronic use of medications/supplements that can potentially affect gut microbiota (i.e. probiotics, anti-inflammatory agents, glucocorticoids, other immune modulating medications, antacids or proton pump inhibitors)
* history of intestinal surgery, inflammatory bowel disease, celiac disease, lactose intolerance, chronic pancreatitis, or other malabsorption disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with underlying cardiomyopathy and having an implantable cardioverter defibrillator for protection from ventricular arrhythmias.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in microbial composition of gut microbiome in study and control groups | 1 year
  Microbial components identified through genetics will be compared between groups.

SECONDARY OUTCOMES:
Change in microbial composition of gut microbiome after successful VT therapy | 1 year
  Microbial components identified through genetics will be compared before and after VT therapy in the high VT burden group.

CONTACTS AND LOCATIONS:
Overall Officials: Ramil Goel, MD, Principal Investigator — Malcolm Randall VAMC
Locations (1):
- Malcolm Randall VA medical center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No